CLINICAL TRIAL: NCT03521284
Title: Health Education : Teaching, Support and Questioning of Young Parents in Maternity
Brief Title: Health Education in the Perinatal Period
Acronym: ESTAQUE
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Other Study IDs: 2017-60
Record Dates: First submitted 2018-03-02; First posted 2018-05-11 (Actual); Last update posted 2018-05-11 (Actual); Status verified 2018-03

CONDITIONS: Postpartum
Keywords: perinatal period
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Mothers with education program during their mat
  Interventions: Other: Parental educational program; Other: Questionnaires
- Mothers without education program during their mat
  Interventions: Other: Questionnaires

INTERVENTIONS:
Other: Parental educational program — Behavior: psychotherapy, life hygiene advice
  Groups: Mothers with education program during their mat
Other: Questionnaires — knowledge questionnaire + parental anxiety questionnaire

SUMMARY:
Health education is now a major public health issue. In the field of perinatal care, the interests involved are the upgrading of the role of mother / father in the health education of their child and the disengagement of inappropriate pediatric consultations and emergency services in front of mothers who " fail know how to ". A recent review of the literature (Cochrane Library) on the effectiveness of parenting programs in the first 2 months of life of the newborn shows that parental education programs focusing on the explanation of newborn rhythms to young parents increased sleeping time to 6 weeks of life or a significant improvement in the prevention of domestic accidents (checking the water temperature and reducing the risk of burning, sleeping in the bed and preventing unexpected sudden death of the infant, position and respect of instructions during transport by car and prevention of road accidents). However, the authors of this meta-analysis concluded that new studies were needed to confirm the results already published.

The main objective of this study is to evaluate the effectiveness of an early parental education program in maternity both in terms of parental acquisitions and their implementation after leaving the service. These parental acquisitions relate, on the one hand, to the care to be given to the newborn child and, on the other hand, on the possible pathologies that he or she could have, and the best action to be taken by the parents to respond to them. The secondary objective is to evaluate the impact of this program on maternal anxiety in this special period of transition to the role of a parent.

It is a prospective, monocentric, comparative, randomized, controlled, open study. The comparison will be made between two experimental groups. The first experimental group corresponds to the mothers who attended the education program during their maternity stay. The second control group corresponds to mothers who did not attend the training. The primary endpoint for measuring this effectiveness is maternal knowledge assessment using knowledge questionnaires that will be completed by mothers before (pre-test) and after (post-test) the educational program in the maternity unit. The secondary endpoints for assessing the primary objective of measuring this effectiveness are the maternal knowledge assessment 1 month after leaving the maternity, using a questionnaire (Recall-Test) and the assessment of the appeal to a medical consultation for the newborn child in the first month of life and the analysis of the relevance of this recourse to the care. The criterion of evaluation of the secondary objective to measure the impact of the educational program on maternal anxiety will be based on questionnaires tested regarding parental anxiety in the perinatal period (STAI-Etat) before and after the educational program.

The investigators believe that this improvement in parental knowledge will have a positive impact on maternal anxiety in the first month of life and will lead to an improvement in the appropriateness of the use of care during the first month of life. If these results are confirmed, this educational program will have a real medico-economic impact (relieving emergency departments and improving the prognosis of newborns with severe pathologies and taken into care earlier by decreasing in parallel the duration of hospitalization).

The impact of these results will allow to promote more widely the health education in the perinatal and neonatal period by generalizing this educational program in other maternities which could be interested. Also, it will allow to propose this educational program in prenatal (within the framework of session of preparation for the birth), after the release from the service, within the framework of structure of health such as the PMI, the community centers and medical structures, even the distribution of these educational program on a larger scale by means of media such as dedicated web site or smartphone applications.

ELIGIBILITY:
Inclusion Criteria:

* Patient giving birth after 37 weeks of amenorrhoea
* Patient giving birth to a newborn child without infectious, malformative or genetic pathology.
* Patient with newborn child hospitalized in Department of Suites de couches, Maternité du pole Femmes-Parents-Enfants, Hopital Nord Marseille

Exclusion Criteria:

* Patient with newborn child requiring home medical care
* Patient donnant naissance à un nouveau-né présentant un faible poids à la naissance

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Young parents in the perinatal and neonatal period
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2018-05 (Estimated); Primary Completion 2018-11 (Estimated); Study Completion 2019-11 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the effectiveness of an early parental education program in maternity | 6 months
  knowledge questionnaires completed by mothers

SECONDARY OUTCOMES:
Evaluation of the impact of the educational program on maternal anxiety | 6 months
  questionnaires tested regarding parental anxiety in the perinatal period (STAI-Etat)

CONTACTS AND LOCATIONS:
Overall Officials: Urielle DESALBRES, Study Director — Assistance Publique Hopitaux De Marseille